CLINICAL TRIAL: NCT02482038
Title: A Single Centre Open Label Pilot Study Measuring Lower Limb Blood Flow in Patients With Venous Leg Ulcers Using the Geko™ T-2 or gekoTM Plus [R-2] Neuromuscular Electro Stimulation Device
Brief Title: Geko Venous Leg Ulcer Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firstkind Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FSK-VLU-001
Record Dates: First submitted 2015-06-23; First posted 2015-06-25 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- geko device (Experimental)
  Interventions: Device: geko

INTERVENTIONS:
Device: geko — neuromuscular electrostimulator

SUMMARY:
This study is designed to look at the effect of the geko device on the circulation in lower limbs of participants with venous leg ulcers.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Intact healthy skin at the site of device application
3. Able to understand the Patient Information Sheet
4. Willing to give informed consent
5. Willing to follow the requirements of the protocol
6. Subjects who had a chronic venous leg ulcer (i.e. CEAP classification of C6 1) greater than 2 cm2 and less than 10 cm in maximum diameter,
7. ABPI of 0.8 or greater

Exclusion Criteria:

1. History of significant haematological disorders or DVT with the preceding six months
2. Pregnant
3. Pacemakers or implantable defibrillators
4. Use of any other neuro-modulation device
5. Current use of TENS in pelvic region, back or legs
6. Use of investigational drug or device within the past 4 weeks that may interfere with this study
7. Recent surgery (such as abdominal, gynaecological, hip or knee replacement)
8. Recent trauma to the lower limbs
9. Size of leg incompatible with the geko™ device.
10. Chronic obesity (BMI > 34)
11. Any medication deemed to be significant by the Investigator
12. Subjects who had an index venous leg ulcer greater in maximum diameter than 10cm in any one dimension
13. Diabetic subjects with advanced small vessel disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Ultra sound measurements of haemodynamics | 10mins

SECONDARY OUTCOMES:
Adverse event rate | 2 hrs
patient rated tolerability | 2 hrs
  A questionnaire has been designed to record the opinion of the patient with regard to the device, in particular how comfortable the device was to wear. The patient will be asked to rate how comfortable the devices are to wear on a scale of 1-5, 1 being very comfortable and 5 being extremely uncomfortable

CONTACTS AND LOCATIONS:
Locations (1):
- Ealing Hospital, Ealing, Middlesex, United Kingdom